CLINICAL TRIAL: NCT00603889
Title: Development of a Skin Test to Detect Immediate-type Hypersensitivity to the Experimental Na-ASP-2 Hookworm Antigen
Brief Title: Development of a Skin Test for the Na-ASP-2 Hookworm Antigen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert B. Sabin Vaccine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SVI-07-02
Record Dates: First submitted 2008-01-17; First posted 2008-01-29 (Estimated); Results first posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-01

CONDITIONS: Hookworm Infection; Allergy
Keywords: Hookworm; Allergy; Vaccine; Skin test
MeSH Terms: conditions — Hookworm Infections; Hypersensitivity; Ancylostomiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Na-ASP-2 Hookworm Antigen Skin Test (Experimental): All participants will have the same number of concentrations of the Na-ASP-2 skin test reagent applied to their arms, using both the prick-puncture and intradermal techniques.
  Interventions: Biological: Na-ASP-2 Skin Test Reagent

INTERVENTIONS:
Biological: Na-ASP-2 Skin Test Reagent — Na-ASP-2 Hookworm Skin Test Reagent, 1-1000 mcg/mL solution

SUMMARY:
Na-ASP-2 is a protein expressed during the larval stage of the N. americanus hookworm life cycle. In a clinical study in previously hookworm-infected adults in Brazil, this protein induced urticarial reactions (rash) in a subset of volunteers. This study will evaluate solutions of varying concentrations of the protein in both a skin prick-puncture and intradermal test that will eventually be used to screen volunteers living in hookworm endemic areas who are being considered as potential participants in vaccine trials, to reduce the potential of inducing allergic reactions in those vaccinated with the Na-ASP-2 Hookworm Vaccine.

DETAILED DESCRIPTION:
* Study site: George Washington University Medical Center
* Number of participants: up to 15
* Study duration: up to 3 months; each participant will undergo a minimum of one screening visit and one study visit.
* Each participant will have both skin prick-puncture and intradermal skin tests applied on the same study day. The prick-puncture and intradermal tests will be applied sequentially to the volar aspects of the participant's forearms:

  1. Skin prick-puncture: four different concentrations of Na-ASP-2 solution (1, 10, 100, and 1000 μg/mL) will be applied simultaneously in duplicate, to the left forearm.
  2. Intradermal: three different concentrations of Na-ASP-2 (10, 100, and 1000 μg/mL) will be injected simultaneously, in duplicate, to the right forearm.
  3. Allergen diluent and histamine solutions will be utilized as the negative and positive controls, respectively, for both the skin prick-puncture and intradermal tests.
  4. Participants will be observed in the study clinic for at least 30 minutes following application of the skin tests, and will be contacted via telephone 2 days following skin testing.
  5. Sizes of the wheal and erythema reactions for each application will be recorded and graded in comparison to the histamine positive control reaction.
* Each participant will have blood collected via venipuncture (a maximum of 25 mL) immediately prior to application of the skin tests, in order to measure antibodies (particularly IgG and IgE) to Na-ASP-2 using an ELISA procedure.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 45 years of age, inclusive.
* Good general health as determined by means of the screening procedure.
* Willingness to participate in the study as evidenced by signing the informed consent document.

Exclusion Criteria:

* History of previous infection with hookworm.
* Prior extensive and continuous travel, work, or residence (> 1 month) in a hookworm-endemic region.
* Pregnancy as determined by a positive urine hCG test (if female).
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history or physical examination.
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
* Participation in an investigational vaccine or drug trial within 14 days of starting this study.
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Known immunodeficiency syndrome.
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study.
* History of a surgical splenectomy.
* Extensive dermatitis precluding skin testing
* Current use of a beta blocker (oral or topical) or anti-histamine medication. A volunteer may participate in the study if they agree to withhold use of an anti-histamine for at least 5 days prior to application of the skin test.
* Use of a tricyclic anti-depressant within the past month.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Parenti, MD, Principal Investigator — GWUMC Medical Faculty Associates
Locations (1):
- GWUMC Clinical Trials Unit, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Fujiwara RT, Bethony J, Bueno LL, Wang Y, Ahn SY, Samuel A, Bottazzi ME, Hotez P, Mendez S. Immunogenicity of the hookworm Na-ASP-2 vaccine candidate: characterization of humoral and cellular responses after vaccination in the Sprague Dawley rat. Hum Vaccin. 2005 May-Jun;1(3):123-8. doi: 10.4161/hv.1.3.1924. Epub 2005 May 20. PMID 17012856
- [Background] Goud GN, Bottazzi ME, Zhan B, Mendez S, Deumic V, Plieskatt J, Liu S, Wang Y, Bueno L, Fujiwara R, Samuel A, Ahn SY, Solanki M, Asojo OA, Wang J, Bethony JM, Loukas A, Roy M, Hotez PJ. Expression of the Necator americanus hookworm larval antigen Na-ASP-2 in Pichia pastoris and purification of the recombinant protein for use in human clinical trials. Vaccine. 2005 Sep 15;23(39):4754-64. doi: 10.1016/j.vaccine.2005.04.040. PMID 16054275
- [Background] Diemert DJ, Bethony JM, Hotez PJ. Hookworm vaccines. Clin Infect Dis. 2008 Jan 15;46(2):282-8. doi: 10.1086/524070. PMID 18171264

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between March and May 2008, primarily by means of advertising the study in and around The George Washington University, where the study site is located.
Period: Overall Study
Arm/Group | Na-ASP-2 Hookworm Antigen Skin Test
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Na-ASP-2 Hookworm Antigen Skin Test
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: 100 Mcg/ml Na-ASP-2 Prick-puncture Skin Test
Description: Mean grade of wheal reaction after 2 applications of the skin test reagent per participant. For each skin test reaction, the grade of the test was determined based on the mean of the longest and orthogonal diameters, which was then compared to the equivalent measurements of a histamine solution positive control that was applied at the same time as the test. Grading was as follows:
  0 no discernible wheal
  1. < ½ histamine diameter
  2. ≥ ½ histamine; < histamine diameter
  3. = size of histamine control ± 1 mm
  4. > histamine diameter; < 2x diameter
  5. ≥ 2x histamine control
Time Frame: 15 minutes after skin test application
Measure: Mean (Full Range); unit: Units on a scale
Groups:
- Na-ASP-2 Hookworm Antigen Skin Test: Application of different concentrations of the Na-ASP-2 antigen skin test reagent as prick-puncture ("scratch test") and intradermal injections, applied to participants' forearms.
Arm/Group | Na-ASP-2 Hookworm Antigen Skin Test
Number analyzed (Participants) | 12
Units on a scale | 0 [0 to 0]

2. Secondary Outcome: 1000 Mcg/ml Na-ASP-2 Prick-puncture Skin Test
Description: as for outcome 1
Time Frame: 15 minutes after skin test application
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Na-ASP-2 Hookworm Antigen Skin Test
Number analyzed (Participants) | 12
units on a scale | 0.21 [0 to 2]

3. Secondary Outcome: 100 Mcg/ml Na-ASP-2 Intradermal Skin Test
Description: as for outcome 1
Time Frame: 15 minutes after skin test application
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Na-ASP-2 Hookworm Antigen Skin Test
Number analyzed (Participants) | 12
units on a scale | 0.17 [0 to 2]

4. Secondary Outcome: 1000 Mcg/ml Na-ASP-2 Intradermal Skin Test
Description: as for outcome 1
Time Frame: 15 minutes after skin test application
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Na-ASP-2 Hookworm Antigen Skin Test
Number analyzed (Participants) | 12
units on a scale | 1.25 [0 to 2]

ADVERSE EVENTS:
Arm/Group | Na-ASP-2 Hookworm Antigen Skin Test
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Na-ASP-2 Hookworm Antigen Skin Test (N=12)
Delayed Skin Test Reaction (Skin and subcutaneous tissue disorders) | 2 (2) — Delayed skin test reaction at site of application of skin test reagent, consisting of erythema, induration, pain, and pruritus. Reactions occurred approximately 1-3 weeks following application of the skin test.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No